CLINICAL TRIAL: NCT01166269
Title: Intralymphatic Specific Immunotherapy - as a New Treatment Form for Grass-pollen Allergic Subjects
Brief Title: Study to Asses Efficacy of Intralymphatic Immunotherapy
Acronym: ILIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Principal Investigator, Professor, Dr. Med Hans-Joergen Malling, Professor Dr. Med., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ILIT
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Allergy
Keywords: grass-pollen allergy
MeSH Terms: conditions — Hypersensitivity | interventions — PHLPVI protein, Phleum pratense

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Grass-Allergen x 6 (Experimental): This arm will receive 6 injections of allergen.
  Interventions: Biological: phleum pratense (grass-allergen)
- grass-allergen x 3 and placebo x 3 (Active Comparator): this arm will receive 3 injections of allergen, and 3 injections of placebo.
  Interventions: Biological: phleum pratense (grass allergen)
- placebo x 6 (Placebo Comparator): this arm will receive 6 injections of placebo.
  Interventions: Other: physiological saline

INTERVENTIONS:
Biological: phleum pratense (grass-allergen) — 6 injections of grass-allergen. Every dose will be 1000 SQ-U.
  Arms: Grass-Allergen x 6
Biological: phleum pratense (grass allergen) — 3 injections of grass-allergen. Every dose will be 1000 SQ-U. Also 3 injections of placebo (physiological saline)
  Arms: grass-allergen x 3 and placebo x 3
Other: physiological saline — 6 injections of placebo (physiological saline)in a lymph node.
  Arms: placebo x 6

SUMMARY:
The purpose of the study is to try a new route for specific immunotherapy (SIT). The current treatment form for SIT is subcutaneously (SCIT), which is a long treatment with up to 50 injections subcutaneously in the upper arm.

The investigators believe that there is additional effect if the allergen is injected directly into the lymph node, since it is here, the allergen presentation is happening. The trial has been performed in Switzerland with significant effect of only three injections of grass-allergen into a lymph node (Clinicaltrials.gov; NCT00470457).

The investigators would like to see what happens if the the dose is doubled, so the patients will receive 6 injections all in all, with the same amount of allergen as the earlier study (1000 SQ-U). Also the outcome measurements is slightly different as the patients will note their symptoms in a diary.

The patients will be divided into three groups using allocation:

1 group with 6 injections of allergen

1 group with 3 injections of allergen and 3 injections of placebo

1 group with 6 injections of placebo. The trial will be double blinded.

ELIGIBILITY:
Inclusion Criteria:

* grass pollen allergy through at least 2 seasons
* positive skin prick test
* positive Specific IgE of at least 2. (CAP)
* Signed informed consent
* for females a negative pregnancy test.

Exclusion Criteria:

* out of age limits
* rhinoconjunctivitis all year round.
* uncontrolled seasonal asthma
* patients treated with steroids continuously or beta-blockers.
* pregnancy and breastfeeding
* HIV, Hepatitis B+c, and other immunological diseases.
* psychiatric disease
* treatment with SCIT or SLIT within the last 5 years
* participation in other clinical trials within the last 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
symptom improvement | 2 seasons. (2 years)
  The patients will fill out a diary during the grasspollen-season before and after treatment. Also they will fill out a form for the general status of the season passed.

SECONDARY OUTCOMES:
Improvement of reactivity of skin prick test and Specific IgE | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joergen Malling, Prof. Dr. Med., Principal Investigator — Copenhagen University Hospital, Gentofte, Denmark
Locations (1):
- Dermato-allergological dept. K, Gentofte Municipality, Hellerup, Denmark